CLINICAL TRIAL: NCT00474058
Title: Phase 3B, Multicenter, Multinational, Double-Blind, Placebo Controlled, 2-Arm Trial to Evaluate the Effect of the 24-Hour Transdermal Delivery of Rotigotine on the Control of Early Morning Motor Function, Sleep Quality, Nocturnal Symptoms, and Non-Motor Symptoms in Subjects With Idiopathic Parkinson's Disease
Brief Title: Randomized Evaluation of the 24-Hour Coverage: Efficacy of Rotigotine
Acronym: RECOVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP0889; EudraCT No.: 2006-006752-35 (Other: EudraCT)
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Results first posted 2010-04-12 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-05

CONDITIONS: Parkinson's Disease
Keywords: rotigotine; Neupro®; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine (Experimental): Rotigotine transdermal patch
  Interventions: Drug: Rotigotine
- Placebo (Placebo Comparator): Placebo transdermal patch
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rotigotine — Rotigotine transdermal patches:
  10cm2 (2mg/24h); 20cm2 (4mg/24h); 30cm2 (6mg/24h); 40cm2 (8mg/24h)
  Optimal dosing: The maximum Rotigotine dose allowed is 16mg/24h
  Other Names: Neupro
  Arms: Rotigotine
Other: Placebo — Placebo transdermal patches
  Arms: Placebo

SUMMARY:
The objective of this trial is to assess the effects of transdermal rotigotine on the control of early morning motor function and sleep disorders compared to placebo in subjects with idiopathic Parkinsons´s disease. In addition, effects of rotigotine on specific nocturnal and non-motor symptoms of Parkinson´s disease will be evaluated.

DETAILED DESCRIPTION:
The objective of this trial is to assess the effects of rotigotine on the control of early morning motor function and sleep disorders compared to placebo in subjects with idiopathic Parkinsons´s disease. In addition, effects of rotigotine on specific nocturnal and non-motor symptoms of Parkinson´s disease will be evaluated.

After a Screening Period of up to 28 days subjects will be hospitalized for two nights. After the second overnight stay, subjects will be randomly assigned either to rotigotine patch or placebo patch. Afterwards patients will be titrated to their optimal dose. After subjects have reached their optimal dose (or the highest dose) they will be maintained on this dose for a certain period. At the end of maintenance the subjects will be hospitalized for two nights. Afterwards the doses will be continuously decreased.

Efficacy will be assessed by application of sleep quality scores, motor examination scores, and scores to evaluate non-motor symptoms of Parkinsons. Safety assessments include adverse events, 12-lead electrocardiograms, blood pressure and heart rate assessments, and laboratory checks.

ELIGIBILITY:
Inclusion Criteria:

* Early and advanced Idiopathic Parkinson Disease with early morning motor impairment

Exclusion Criteria:

* Atypical Parkinsonian syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2007-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (46):
- United States (7):
  - Reseda, California
  - Ventura, California
  - St. Petersburg, Florida
  - Salisbury, North Carolina
  - Winston_Salem, North Carolina
  - Warwick, Rhode Island
  - Houston, Texas
- Australia (3):
  - Concord, New South Wales
  - Adelaide, South Australia
  - Fitzroy
- Innsbruck, Austria
- Finland (2):
  - Hyvinkää
  - Oulu
- Germany (7):
  - Berlin
  - Dresden
  - Kassel
  - Leipzig
  - Marburg
  - Naumburg
  - Ulm
- Hungary (4):
  - Budapest
  - Debrecen
  - Nyíregyháza
  - Zalaegerszeg
- Italy (3):
  - Chieti
  - Milan
  - Torino
- New Zealand (2):
  - Christchurch
  - Wellington
- Poland (6):
  - Gdansk
  - Krakow
  - Lublin
  - Olsztyn
  - Szczecin
  - Warsaw
- South Africa (5):
  - Cape Town
  - Capetown
  - Johannesburg
  - Pretoria/Gauteng
  - Tygerberg
- Spain (2):
  - Barcelona
  - Madrid
- United Kingdom (4):
  - Bristol
  - Lancashire
  - Liverpool
  - London

REFERENCES:
- [Result] Ghys L, Surmann E, Whitesides J, Boroojerdi B. Effect of rotigotine on sleep and quality of life in Parkinson's disease patients: post hoc analysis of RECOVER patients who were symptomatic at baseline. Expert Opin Pharmacother. 2011 Sep;12(13):1985-98. doi: 10.1517/14656566.2011.604031. Epub 2011 Jul 27. PMID 21790503
- [Derived] Kassubek J, Chaudhuri KR, Zesiewicz T, Surmann E, Boroojerdi B, Moran K, Ghys L, Trenkwalder C. Rotigotine transdermal system and evaluation of pain in patients with Parkinson's disease: a post hoc analysis of the RECOVER study. BMC Neurol. 2014 Mar 6;14:42. doi: 10.1186/1471-2377-14-42. PMID 24602411
- [Derived] Swick TJ, Friedman JH, Chaudhuri KR, Surmann E, Boroojerdi B, Moran K, Ghys L, Trenkwalder C. Associations between severity of motor function and nonmotor symptoms in Parkinson's disease: a post hoc analysis of the RECOVER Study. Eur Neurol. 2014;71(3-4):140-7. doi: 10.1159/000355019. Epub 2014 Jan 21. PMID 24457253
- [Derived] Trenkwalder C, Kies B, Rudzinska M, Fine J, Nikl J, Honczarenko K, Dioszeghy P, Hill D, Anderson T, Myllyla V, Kassubek J, Steiger M, Zucconi M, Tolosa E, Poewe W, Surmann E, Whitesides J, Boroojerdi B, Chaudhuri KR; Recover Study Group. Rotigotine effects on early morning motor function and sleep in Parkinson's disease: a double-blind, randomized, placebo-controlled study (RECOVER). Mov Disord. 2011 Jan;26(1):90-9. doi: 10.1002/mds.23441. Epub 2010 Nov 18. PMID 21322021
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 333 subjects were enrolled in this trial and comprised the Enrolled Set (ES). 287 subjects were randomized and all of them received at least 1 dose of trial medication, so they all belong to the Safety Set (SS). 267 subjects belong to the Full Analysis Set (FAS).
Pre-assignment Details: Participant Flow shows all 287 subjects who has been enrolled and randomized. Baseline Characteristics are described for the Full Analysis Set (FAS).
Period: Overall Study
Arm/Group | Rotigotine | Placebo
Started | 190 | 97
Completed | 166 | 80
Not Completed | 24 | 17
Not completed — Adverse Event | 11 | 6
Not completed — Lack of Efficacy | 0 | 4
Not completed — Withdrawal by Subject | 11 | 7
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotigotine | Placebo | Total
Number analyzed (Participants) | 178 | 89 | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 87 | 40 | 127
  >=65 years | 91 | 49 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.4) | 64.5 (10.4) | 64.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 31 | 92
  Male | 117 | 58 | 175
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 164 | 79 | 243
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 8 | 19
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/ m^2] | 26.676 (4.164) | 26.645 (4.569) | 26.665 (4.295)
Height [Mean (Standard Deviation); unit: cm] | 169.04 (9.11) | 170.73 (9.27) | 169.60 (9.18)
Weight [Mean (Standard Deviation); unit: kg] | 76.6 (15.1) | 78.0 (16.2) | 77.1 (15.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Early Morning UPDRS Part III Score
Description: The Unified Parkinson´s Disease Rating Scale Part III score is an accepted and validated sumscore of 14 items for the assessment of motor function in Parkinson´s disease. Each of the 14 items in the UPDRS part III is measured on a scale of 0 to 4, where 0 is normal and 4 represents severe abnormalities.
Time Frame: From baseline to end of maintenance (after 4 weeks maintenance)
Population: Full Analysis Set (FAS) with Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 178 | 89
units on a scale | -7.0 (7.6) | -3.9 (7.3)
Statistical Analysis 1: Comparison: Rotigotine vs Placebo; Analyses of covariance were performed for the efficacy variables with treatment and (pooled) sites as factors, and baseline value as covariate. Least square means (LS means) for treatment effect were calculated and differences between rotigotine and placebo were presented with 95% confidence intervals (CIs) and p- values; Test type: Superiority or Other; p = 0.0002, ANCOVA — No p-value adjustment was necessary, since a multiple test procedure in a hierarchical sequentially rejective manner for the primary variable was applied; Mean Difference (Final Values) = -3.55, 95% CI [-5.37 to -1.73]

2. Primary Outcome: Change in Parkinson's Disease Sleep Scale (PDSS)
Description: The Parkinson´s Disease Sleep Scale (PDSS) is a questionnaire with 15 questions to assess sleep and nocturnal disability in Parkinson´s disease. The item- scores can range between 0= never and 4= very often. The PDSS score is a sumscore of all 15 questions.
Time Frame: From baseline to end of maintenance (after 4 weeks maintenance)
Population: Full Analysis Set (FAS) with Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 178 | 89
units on a scale | -5.9 (7.6) | -1.9 (8.2)
Statistical Analysis 1: Comparison: Rotigotine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — No p-value adjustment was necessary, since a multiple testing in a hierarchical sequentially rejective manner for the primary variable was applied; Mean Difference (Final Values) = -4.26, 95% CI [-6.08 to -2.45]

3. Secondary Outcome: Change in Nocturnal Akinesia, Dystonia, and Cramps Score (NADCS)
Description: Subjects were asked to assess nocturnal akinesia, dystonia and cramps, using an ordinal severity scale. While a score of 0= normal and 4= maximal severity, subjects could also rate their symptoms with values of 0.5, 1.5, 2.5, 3.5. The nocturnal akinesia score was used to evaluate motor performance while the dystonia and cramps scores were used to evaluate sleep.
Time Frame: From baseline to end of maintenance (after 4 weeks maintenance)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 163 | 78
units on a scale | -1.3 (1.8) | -0.9 (2.1)
Statistical Analysis 1: Comparison: Rotigotine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0301, ANCOVA; Mean Difference (Final Values) = -0.41, 95% CI [-0.79 to -0.04]

4. Secondary Outcome: Change in Number of Nocturias
Description: Nocturia is the need to get up during the night and interrupt sleep in order to urinate. It is a typical nocturnal symptom of Parkinson´s disease. The change from baseline in number of nocturias was used to evaluate improvements in sleep disorders.
Time Frame: From baseline to end of maintenance (after 4 weeks maintenance)
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: nocturias
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 161 | 78
nocturias | -0.3 (1.3) | -0.2 (1.1)
Statistical Analysis 1: Comparison: Rotigotine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8842, ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI [-0.29 to 0.25]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to 22 weeks from Visit 1 to the Safety Follow- Up Visit.
Description: Serious and non- serious Adverse Events (AEs) refer to the Safety Set (SS). The SS includes all subjects who are randomized and received at least one dose of trial medication.
Arm/Group | Rotigotine | Placebo
Serious Adverse Events (participants affected / at risk) | 10/191 | 5/96
Other Adverse Events (participants affected / at risk) | 70/191 | 21/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=191) | Placebo (N=96)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep attacks (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=191) | Placebo (N=96)
Nausea (Gastrointestinal disorders) | 41 (54) | 9 (14)
Dizziness (Nervous system disorders) | 20 (27) | 6 (6)
Headache (Nervous system disorders) | 13 (14) | 5 (5)
Dyskinesia (Nervous system disorders) | 15 (16) | 4 (4)

LIMITATIONS AND CAVEATS:
During the course of the trial, the manufacturing process for rotigotine was changed. At that time, the expiry date for trial medication was Apr 2009, recruitment for SP889 had to be stopped effective on 17 Nov 2008.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome."